CLINICAL TRIAL: NCT03307928
Title: Can Obstructive Sleep Apnea Impair Cardiorespiratory Responses to Aerobic Exercise in Hypertensive Elderly?
Brief Title: Cardiorespiratory Responses to Exercise in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Bruno Teixeira Barbosa, Assistant Professor, Federal University of Paraíba
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 48423815.1.0000.5188
Record Dates: First submitted 2017-03-22; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Obstructive Sleep Apnea Syndrome; Aged; Hypertension; Oxygen Consumption; Exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: The participants were divided into two groups: (1) hypertension without OSA (NO-OSA group; AHI < 5 events/h; n = 15) and (2) hypertension with OSA (OSA group: AHI ≥ 15 events/h; n = 13).
Who Masked: Participant, Investigator
Masking Description: The investigator did not have access to the exams that the volunteers realized, either they have access to what they were doing or the order of the exams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiopulmonary Exercise Test Protocol (Experimental): All subjects performed an incremental cardiopulmonary exercise test (CPET) to maximum exercise tolerance. All the procedures were performed in agreement with the American Thoracic Society/American College of Chest Physicians guidelines for cycle ergometer tests.
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Test Protocol; Diagnostic Test: Polysomnography Assessment
- Polysomnography Assessment (Experimental): All hypertensive subjects were submitted to a polysomnography exam to diagnose OSA. The OSA diagnose was confirmed by the apnea/hypopnea index (AHI) and classified as follows: AHI < 5 events/h, absence of OSA; 5 ≤ AHI ≤ 15 events/h, low OSA; 15 ≤ AHI ≤ 30 events/h, moderate OSA; AHI > 30 events/h, severe OSA.
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Test Protocol; Diagnostic Test: Polysomnography Assessment

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Test Protocol — The CPET was performed in a cycle ergometer with electromagnetic braking using an Inbrasport (Inbrasport, Porto Alegre, Rio Grande do Sul, Brazil). Following a 5-min warm-up against no resistance (0 W), the work rate was increased using a ramp protocol (5-10 W.min-1) until maximum exercise tolerance. Verbal encouragements were given during the CPET to ensure maximal effort.
Diagnostic Test: Polysomnography Assessment — The polysomnography assessment was carried out during an entire night of sleep in the participant's residence with no use of sedatives. The variables were monitored by an Embletta portable respiratory monitor (Embla, Embletta® Gold, EUA), previously validated, and in agreement with manufacturer's instructions. The Embletta monitor was capable to monitor continuously the pulse oximetry, to detect respiratory efforts, to measure the airflow, and to record snoring episodes. Additionally, HR was continually measured by the analysis of pulse waves by oximetry. Finally, brain and muscle activities were monitored by electrodes and oxygen desaturation (O2D) was defined as the amount of reduction in O2S in 4%/h.

SUMMARY:
Elderly have a high prevalence to systemic arterial hypertension (SAH) and obstructive sleep apnea (OSA). Both comorbidities are closely associated and inflict injury cardiorespiratory capacity. To assess cardiorespiratory responses to the cardiopulmonary exercise test (CPET) among hypertensive elderly with OSA. We enrolled 25 elderly hypertensive in two different groups: without OSA (No-OSA: Apnea/Hypopnea Index (AHI) < 5 events/h; n = 15) and with OSA (OSA: AHI ≥ 15 events/h; n = 13). All subjects underwent a CPET and polysomnographic assessments. After normality and homogeneity evaluations, independent t test and pearson's correlation were performed. The significance level was p ≤ 0.05.

DETAILED DESCRIPTION:
The sample was randomly recruited from the Lauro Wanderley University Hospital and older people living together centers located in João Pessoa/PB (Brazil). All subjects were submitted to anthropometric assessments (body mass index, neck circumference, hip circumference and waist circumference), polysomnography, echocardiography, cardiopulmonary exercise test (CPET). Moreover, they were submitted to a sleep quality questionnaire (Pittsburgh Sleep Quality Index).

Cardiopulmonary Exercise Test Protocol All subjects performed an incremental cardiopulmonary exercise test (CPET) of maximum exercise tolerance. All procedures were performed in agreement with the guidelines of the American Thoracic Society/American College of Chest Physicians for cycle ergometer tests. The CPET was performed on an Inbrasport CG-04 cycle ergometer (Inbrasport, Porto Alegre, Rio Grande do Sul, Brazil) with electromagnetic braking. Subjects performed a 5-min warm-up with no resistance (0 W), then the activity rate was increased using a ramp protocol (5-10 W.min-1) until maximum exercise tolerance. Verbal encouragements were given during the CPET to ensure maximal effort.

Pulmonary gas exchange variables (VO2, VCO2, minute ventilation [VE], oxygen pulse (O2Pu), respiratory quotient (R), ventilatory efficiency index (VE/VCO2slope), cardiovascular function index (ΔHR/ΔVO2), deviation from oxygen consumption efficiency (OUES), metabolic efficiency index (VO2/ΔWR), blood pressure (BP), heart rate (HR) recovery at first (HRR1) and second (HRR2) minutes were measured breath-by-breath with an on-line gas expiration analysis system (VO2000, MedGraphics, St. Paul, Minnesota, USA). Peak values were established by the highest values achieved during effort.

Polysomnography Assessment All hypertensive subjects were submitted to a polysomnography exam to diagnose OSA. OSA diagnosis was confirmed by the apnea/hypopnea index (AHI) and classified as follows: AHI < 5 events/h, absence of OSA; 5 ≤ AHI ≤ 15 events/h, low OSA; 15 ≤ AHI ≤ 30 events/h, moderate OSA; AHI > 30 events/h, severe OSA.

The assessment was carried out during an entire night of sleep in the participant's residence without the use of sedatives. The variables were monitored by an Embletta portable respiratory monitor (Embla, Embletta® Gold, EUA), previously validated and in agreement with manufacturer's instructions. The Embletta monitor is capable to continuously monitor pulse oximetry, to detect respiratory efforts, to measure the airflow, and to record snoring episodes. Additionally, HR was continually measured by the analysis of pulse waves by oximetry. Finally, brain and muscle activities were monitored by electrodes, and oxygen desaturation (O2D) was defined as the amount of reduction in O2S at 4%/h.

Echocardiography All subjects performed the two-dimensional color Doppler echocardiogram (iE33® - Philips Electronics, Netherlands) before the CPET. Final systolic and diastolic diameters of the left ventricle and the diastolic thickness of the posterior wall of the left ventricle were measured from the short-axis view, and ejection fraction was obtained from these measures. This exam was conducted by an experienced cardiologist, who was blinded to group allocation.

Sleep Quality The subjective sleep quality was assessed by the Pittsburgh Sleep Quality Index, which consists of 19 questions grouped into 7 different components (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disorders, use of medications, and diurnal dysfunction). The classifications depended upon the scores reached in each question (from 0 to 3); ranging from 0 - 4: good subjective sleep quality; 5 - 10: bad subjective sleep quality; and 11 or higher: indicates the presence of at least one sleep disorder.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in stage I or II of systemic hypertension without use of beta-blockers, eutrophics, non-smokers (< 6 months), with no diabetes, or any respiratory or cardiovascular disease and considered irregularly active [15] were enrolled in this study.

Exclusion Criteria:

* Those with diabetes or any respiratory or cardiovascular disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | A entire night sleep, an average of 8 yours.
  The OSA diagnose was confirmed by the apnea/hypopnea index (AHI) and classified as follows: AHI < 5 events/h, absence of OSA; 5 ≤ AHI ≤ 15 events/h, low OSA; 15 ≤ AHI ≤ 30 events/h, moderate OSA; AHI > 30 events/h, severe OSA.

SECONDARY OUTCOMES:
Oxygen Consumption | A entire procedure (approximately 10 minutes)
  Following a 5-min warm-up against no resistance (0 W), the work rate was increased using a ramp protocol (5-10 W.min-1) until maximum exercise tolerance. Verbal encouragements were given during the CPET to ensure maximal effort.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Barbosa, Master, Principal Investigator — Centro Universitário de João Pessoa
Locations (1):
- Bruno Teixeira Barbosa, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No